CLINICAL TRIAL: NCT06547619
Title: Role of ET-1, Physical Activity, and Sedentary Behavior in Microvascular Dysfunction Following GDM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202405270
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes; Endothelial Dysfunction; Physical Inactivity
MeSH Terms: conditions — Diabetes, Gestational; Sedentary Behavior | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- local lactated Ringer's perfusion (Placebo Comparator): lactated Ringer's is perfused through the microdialysis fiber to serve as the vehicle control
  Interventions: Drug: Insulin aspart
- local BQ-788 and BQ-123 perfusion (Experimental): local ET-1 inhibitors perfused through the microdialysis fiber to serve as the experimental treatment
  Interventions: Drug: Insulin aspart
- local L-NAME perfusion (Experimental): local L-NAME is perfused through the microdialysis fiber to inhibit nitric oxide synthase
  Interventions: Drug: Insulin aspart
- local BQ-788 + BQ-123 + L-NAME perfusion (Experimental): local ET-1 inhibitors and L-NAME are perfused through the microdialysis fiber to inhibit nitric oxide synthase during the experimental treatment
  Interventions: Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin aspart — insulin aspart is perfused at 5 ascending concentrations (10^-8M - 10^-4 M) for 10 minutes each

SUMMARY:
Women with a history of gestational diabetes mellitus (GDM) are at a 2-fold greater risk for the development of overt cardiovascular disease (CVD) following the effected pregnancy. While subsequent development of type II diabetes elevates this risk, prior GDM is an independent risk factor for CVD morbidity, particularly, within the first decade postpartum. GDM is associated with impaired endothelial function during pregnancy and decrements in macro- and microvascular function persist postpartum, despite the remission of insulin resistance following delivery. Collectively, while the association between GDM and elevated lifetime CVD risk is clear, and available evidence demonstrates a link between GDM and vascular dysfunction in the decade following pregnancy, the mechanisms mediating this persistent dysfunction remain unexamined.

The purpose of this investigation is to examine the role of endothelin-1, a potent vasoconstrictor, in aberrant microvascular function in otherwise healthy women with a history of GDM and to identify whether this mechanism is influenced by physical activity and sedentary behavior.

ELIGIBILITY:
INCLUSION CRITERIA

* history of pregnancy within 5 years of the study visit
* had healthy pregnancy OR had gestational diabetes diagnosed by their obstetrician and confirmed according to the American College of Obstetricians and Gynecologists criteria for gestational diabetes.

EXCLUSION CRITERIA

* skin diseases,
* current tobacco or electronic cigarette/vape pen use,
* diagnosed or suspected hepatic or metabolic disease including diabetes,
* statin or other cholesterol-lowering medication,
* current antihypertensive medication,
* history of preeclampsia or gestational hypertension
* current hypertension,
* current pregnancy,
* body mass index <18.5 kg/m2,
* allergy to materials used during the experiment.(e.g. latex), known allergies to study drugs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
amount of microvascular insulin-mediated dilation | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator responses to insulin perfusion in lactated Ringer's, BQ 788 and BQ-123, and L-NAME treated microdialysis sites

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States